CLINICAL TRIAL: NCT02134548
Title: Determination of Estimated Sensitivity for Chagas Detect Plus Rapid Tests
Brief Title: Sensitivity Study of Diagnostic for Detection of Chagas Infection
Status: Completed | Type: Observational
Sponsor: InBios International, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: DSC0226
Record Dates: First submitted 2014-05-07; First posted 2014-05-09 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2015-12

CONDITIONS: Infectious Diseases
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Observational Model: Case-Only
Biospecimen Retention: Samples Without DNA — serum

SUMMARY:
This study is a multi-site trial assessing the sensitivity of Chagas Detect™ Plus rapid test versus standard reference tests (e.g. IFA, IHA, RIPA) for Chagas diagnosis.

The Chagas Detect™ Plus rapid test serves as an aid in the clinical laboratory diagnosis of Chagas infection in patients. This test is intended to be used on human whole blood or serum samples. Chagas Detect™ Plus results (positive or negative) must be confirmed by testing with a reference standard test.

Subjects will be patients at clinical sites located in Chagas-endemic areas. After informed consent is obtained and the subject is screened for eligibility, 2 diagnostic samples will be collected. One is blood from finger prick, and the other is blood from venous puncture (drawn from vein in arm).

Rapid tests and reference tests will be performed by different operators who are laboratory staff members. These staff members, blinded to each other's results, will evaluate the samples from each method independently.

ELIGIBILITY:
Inclusion Criteria:

* All age groups and both sexes for archive samples, adults only and both sexes for prospective samples.
* Samples collected from subjects living in T. cruzi endemic regions.
* Information must be available about symptoms, age, and sex of patient from which samples are collected.
* The location of sample collection must be recorded.

Exclusion Criteria:

* Archived samples with linked personal identifiers or any sample for which personal information can be discovered.
* Prospective samples from nursing home residents; inmates/subjects in police custody; participants who are unable to understand verbal or written local language in which a certified translation of the informed consent is available, or requires a Legal Authorized Representative (LAR) for consent.
* Subject serum specimens that have undergone more than 2 freeze-thaw cycles or that have not been stored frozen.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Human males and females of varying ages and geographical locations where Chagas infection is endemic. We will use retrospective (archived) and prospective human serum and blood samples.
  Retrospective (archived) serum samples are not collected specifically for this study and are not individually identifiable to the Investigators. These samples will fall under the category of "leftover" specimens as described by FDA guidance.
  Prospective whole blood samples will be collected in compliance with human subject protection. The first sample will be collected from finger prick; the second sample will be collected from venous puncture.
Sampling Method: Probability Sample
Enrollment: 1601 (Actual)
Dates: Start 2013-06; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
number of subjects with positive result | 1 day

CONTACTS AND LOCATIONS:
Locations (2):
- Universidad Catolica Boliviana San Pablo, Unidad Academica Santa Cruz, (Cei), Santa Cruz, Bolivia
- Laboratorio SANALAB, Santiago, Chile